CLINICAL TRIAL: NCT06748014
Title: The Efficacy of Aescin in Combination With Micronized Purified Flavonoid Fraction (MPFF) in the Control of Bleeding and Prevent Recurrence of Acute Internal Hemorrhoids, A Randomized Controlled Trial, A Pilot Study
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Witcha Vipudhamorn, MD, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUR-2567-0485
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Hemorrhoid
Keywords: hemorrhoid; MPFF; Asecin
MeSH Terms: conditions — Hemorrhoids | interventions — Escin; horse chestnut seed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient and assessor doctor dont know what medication the patient recieved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPFF + Placebo (Placebo Comparator): Patient will recived MPFF 3000 mg for 7 day then 1000 mg for 2 month + placebo
  Interventions: Drug: MPFF
- MPFF + Aescin (Active Comparator): Patient will recived MPFF 3000 mg for 7 day then 1000 mg for 2 month + Aescin 60 mg for 2 month
  Interventions: Drug: Aescin in Horse Chestnut; Drug: MPFF

INTERVENTIONS:
Drug: Aescin in Horse Chestnut — Patient will recived MPFF 3000 mg for 7 day then 1000 mg for 2 month + Aescin 60 mg for 2 month
  Arms: MPFF + Aescin
Drug: MPFF — MPFF 3000 mg 7 day then 1000 mg 2 months

SUMMARY:
Hemorrhoidal disease, characterized by symptomatic enlargement and distal displacement of anal cushions, has been a subject of recognition and management for centuries. The etymology of "hemorrhoid" is traced back to the Greek words haima (blood) and rhoos (flow). Prevalent in over 20% of the population across various life stages, this anorectal condition impacts both genders. The multifaceted development of the disease incorporates theories encompassing abnormal dilation of hemorrhoidal plexuses, distension of arteriovenous anastomoses, prolapse of anal pads, and a myriad of genetic, anatomical, dietary, and lifestyle factors. Manifestations range from venous distension to bleeding and thrombosis, with classification based on location (internal/external/combined) and degree of prolapse (grade 1-4).

Upon comprehensive history-taking and examinations, including digital rectal and proctoscope assessments, a definitive diagnosis is established, leading to the treatment phase. Although outpatient procedures demonstrate efficacy, patients may persist with pain and discomfort. Medical intervention assumes significance for stages 1 and 2, incorporating approaches such as rubber-band ligation, injection sclerotherapy, and dietary modifications. Micronized Purified Flavonoid Fraction (MPFF), integral to hemorrhoid treatment, has been scrutinized for its ability to mitigate pathogenic processes culminating in acute bleeding[8]. The stagnation of blood in vascular plexuses prompts an inflammatory response, activating white cells and increasing vessel wall permeability. MPFF's flavonoid compounds are posited to alleviate bleeding by augmenting venous tone, reducing stasis, inhibiting inflammatory mediators, and enhancing lymphatic drainage. Multiple trials substantiate MPFF's efficacy in ceasing bleeding, alleviating symptoms, and preventing hemorrhoid relapse. A recent randomized controlled trial shows that MPFF can cease bleeding hemorrhoids in 3 to 4 days.

Aescin, a saponin mixture found in Aesculus hippocastanum (horse chestnut). The primary active component, β-aescin, contributes to the plant's medicinal attributes. Experimental investigations in animal models underscore its anti-edematous, anti-inflammatory, and venotonic properties, attributed to molecular mechanisms facilitating ion entry into channels and elevating venous tension. In the past, we used aescin for hemorrhoid treatment benefit in reducing mass effect with control bleeding postoperative hemorrhoidectomy. Based on our previous project (SUR-2567-0150), the combination of aescin with MPFF has demonstrated significant efficacy in stopping bleeding and reducing the mass effect in Grade 1 and 2 hemorrhoids. We aim to study the long-term effects of this combination over 1, 3, and 6 months. This study seeks to provide valuable insights that could inform and refine therapeutic strategies for managing hemorrhoids, ultimately improving patient outcomes

DETAILED DESCRIPTION:
Hemorrhoidal disease, characterized by symptomatic enlargement and distal displacement of anal cushions, has been a subject of recognition and management for centuries. The etymology of "hemorrhoid" is traced back to the Greek words haima (blood) and rhoos (flow). Prevalent in over 20% of the population across various life stages, this anorectal condition impacts both genders. The multifaceted development of the disease incorporates theories encompassing abnormal dilation of hemorrhoidal plexuses, distension of arteriovenous anastomoses, prolapse of anal pads, and a myriad of genetic, anatomical, dietary, and lifestyle factors. Manifestations range from venous distension to bleeding and thrombosis, with classification based on location (internal/external/combined) and degree of prolapse (grade 1-4).

Upon comprehensive history-taking and examinations, including digital rectal and proctoscope assessments, a definitive diagnosis is established, leading to the treatment phase. Although outpatient procedures demonstrate efficacy, patients may persist with pain and discomfort. Medical intervention assumes significance for stages 1 and 2, incorporating approaches such as rubber-band ligation, injection sclerotherapy, and dietary modifications. Micronized Purified Flavonoid Fraction (MPFF), integral to hemorrhoid treatment, has been scrutinized for its ability to mitigate pathogenic processes culminating in acute bleeding[8]. The stagnation of blood in vascular plexuses prompts an inflammatory response, activating white cells and increasing vessel wall permeability. MPFF's flavonoid compounds are posited to alleviate bleeding by augmenting venous tone, reducing stasis, inhibiting inflammatory mediators, and enhancing lymphatic drainage. Multiple trials substantiate MPFF's efficacy in ceasing bleeding, alleviating symptoms, and preventing hemorrhoid relapse. A recent randomized controlled trial shows that MPFF can cease bleeding hemorrhoids in 3 to 4 days.

Aescin, a saponin mixture found in Aesculus hippocastanum (horse chestnut). The primary active component, β-aescin, contributes to the plant's medicinal attributes. Experimental investigations in animal models underscore its anti-edematous, anti-inflammatory, and venotonic properties, attributed to molecular mechanisms facilitating ion entry into channels and elevating venous tension. In the past, we used aescin for hemorrhoid treatment benefit in reducing mass effect with control bleeding postoperative hemorrhoidectomy. Based on our previous project (SUR-2567-0150), the combination of aescin with MPFF has demonstrated significant efficacy in stopping bleeding and reducing the mass effect in Grade 1 and 2 hemorrhoids. We aim to study the long-term effects of this combination over 1, 3, and 6 months. This study seeks to provide valuable insights that could inform and refine therapeutic strategies for managing hemorrhoids, ultimately improving patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* Acute active bleeding hemorrhoid grade 1 and 2 with in 7 days
* Age over 20 years
* In patients aged over 50 years, it is imperative to confirm the absence of any alternative causes of bleeding through a colonoscopy
* Can follow up in 6 months

Exclusion Criteria:

* Bleeding disorder
* History of colorectal cancer, inflammatory bowel disease, portal hypertension, chronic kidney disease grade 3 or over
* Patient required other treatment such as hemorrhoidectomy or RBL
* Patient who received antiplatelet or anticoagulant
* Physical exam reveals anal fissure
* Pregnancy
* Any psychotic disorder
* Refuse to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of hemorrhoid | 6 months
  Present of bleeding or protuding mass in1 3 6 month

SECONDARY OUTCOMES:
Stop bleeding in acute phase | 7 day
  Compare efficacy of bleeding cessation in 7 day

CONTACTS AND LOCATIONS:
Overall Officials: WITCHA VIPUDHAMORN, MD, Principal Investigator — Division of Colorectal Surgery, Department of Surgery, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand
Locations (1):
- Chiangmai university, Chiang Mai, Maung, Thailand

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 6 months
Access Criteria: contact via email